CLINICAL TRIAL: NCT03704987
Title: Skeletal Health of Klinefelter Patients is Not so Bad
Brief Title: Skeletal Health of Klinefelter Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Md, Assoc. Prof., TC Erciyes University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2017/33
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Osteoporosis
Keywords: Klinefelter; Osteoporosis; dual-energy X-ray absorptiometry
MeSH Terms: conditions — Osteoporosis; Klinefelter Syndrome | interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: To compare bone mineral density of klinefelter patients and normal population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Klinefelter (Active Comparator): Male patients followed with the diagnosis of klinefelter
  Interventions: Diagnostic Test: dual-energy X-ray absorptiometry
- Control (Active Comparator): healthy male subjects
  Interventions: Diagnostic Test: dual-energy X-ray absorptiometry

INTERVENTIONS:
Diagnostic Test: dual-energy X-ray absorptiometry — dual-energy X-ray absorptiometry

SUMMARY:
This study compared the bone health of KS patients who were actively monitored in our clinic by dual-energy X-ray absorptiometry (DXA) with that of a control group of healthy volunteers.

DETAILED DESCRIPTION:
Klinefelter syndrome (KS) is the most common chromosome number abnormality of men, occurring in 1/500 to 1/1000 live births . It was first described in 1942 as an endocrine disorder characterised by small, hard testicles androgen deficiency, gynaecomastia and increased follicle stimulating hormone (FSH). Osteoporosis is a progressive bone remodelling disorder in which bone loss exceeds bone formation. The resulting micro-architectural defects and bone fragility are associated with increased fracture risk and mortality. In KS, testosterone deficiency is associated with decreased bone mass and low bone mineral density (BMD) , and a positive correlation of total serum testosterone and BMD has been reported . There are some exceptions ; however, most studies have reported that KS increases the risk of osteopenia and osteoporosis compared with age-matched control groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of klinefelter

Exclusion Criteria:

* klinefelter subjects with a history of hip or waist surgery or trauma
* for control group with known bone disease, unknown fertility hypogonadism findings on physical examination (e.g. low testicular volume or abnormal body hair), known hypogonadism, previous androgen replacement therapy any drug therapy affecting bone metabolism

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male patiens
Enrollment: 247 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
BMD | T score obtained from dual-energy X-ray absorptiometry through study completion, an average of 2 years
  bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Demirtas, MD, Principal Investigator — Erciyes University Faculty of Medicine
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paduch DA, Fine RG, Bolyakov A, Kiper J. New concepts in Klinefelter syndrome. Curr Opin Urol. 2008 Nov;18(6):621-7. doi: 10.1097/MOU.0b013e32831367c7. PMID 18832949
- [Background] Manolagas SC. Birth and death of bone cells: basic regulatory mechanisms and implications for the pathogenesis and treatment of osteoporosis. Endocr Rev. 2000 Apr;21(2):115-37. doi: 10.1210/edrv.21.2.0395. PMID 10782361
- [Background] Haentjens P, Magaziner J, Colon-Emeric CS, Vanderschueren D, Milisen K, Velkeniers B, Boonen S. Meta-analysis: excess mortality after hip fracture among older women and men. Ann Intern Med. 2010 Mar 16;152(6):380-90. doi: 10.7326/0003-4819-152-6-201003160-00008. PMID 20231569
- [Background] Center JR, Nguyen TV, Schneider D, Sambrook PN, Eisman JA. Mortality after all major types of osteoporotic fracture in men and women: an observational study. Lancet. 1999 Mar 13;353(9156):878-82. doi: 10.1016/S0140-6736(98)09075-8. PMID 10093980
- [Background] Maravic M, Taupin P, Landais P, Roux C. Decrease of inpatient mortality for hip fracture in France. Joint Bone Spine. 2011 Oct;78(5):506-9. doi: 10.1016/j.jbspin.2010.11.006. Epub 2010 Dec 22. PMID 21183376
- [Background] Liu H, Paige NM, Goldzweig CL, Wong E, Zhou A, Suttorp MJ, Munjas B, Orwoll E, Shekelle P. Screening for osteoporosis in men: a systematic review for an American College of Physicians guideline. Ann Intern Med. 2008 May 6;148(9):685-701. doi: 10.7326/0003-4819-148-9-200805060-00009. PMID 18458282
- [Background] Ferlin A, Schipilliti M, Di Mambro A, Vinanzi C, Foresta C. Osteoporosis in Klinefelter's syndrome. Mol Hum Reprod. 2010 Jun;16(6):402-10. doi: 10.1093/molehr/gaq026. Epub 2010 Mar 27. PMID 20348548
- [Background] Eulry F, Bauduceau B, Lechevalier D, Magnin J, Flageat J, Gautier D. [Early spinal bone loss in Klinefelter syndrome. X-ray computed tomographic evaluation in 16 cases]. Rev Rhum Ed Fr. 1993 Apr;60(4):287-91. French. PMID 8167626
- [Background] Choi HR, Lim SK, Lee MS. Site-specific effect of testosterone on bone mineral density in male hypogonadism. J Korean Med Sci. 1995 Dec;10(6):431-5. doi: 10.3346/jkms.1995.10.6.431. PMID 8924228
- [Background] Foresta C, Ruzza G, Mioni R, Meneghello A, Baccichetti C. Testosterone and bone loss in Klinefelter syndrome. Horm Metab Res. 1983 Jan;15(1):56-7. doi: 10.1055/s-2007-1018630. No abstract available. PMID 6832705
- [Background] Luisetto G, Mastrogiacomo I, Bonanni G, Pozzan G, Botteon S, Tizian L, Galuppo P. Bone mass and mineral metabolism in Klinefelter's syndrome. Osteoporos Int. 1995;5(6):455-61. doi: 10.1007/BF01626608. PMID 8695968
- [Background] Hieronimus S, Lussiez V, Le Duff F, Ferrari P, Bstandig B, Fenichel P. Klinefelter's syndrome and bone mineral density: is osteoporosis a constant feature? Ann Endocrinol (Paris). 2011 Feb;72(1):14-8. doi: 10.1016/j.ando.2010.10.002. Epub 2010 Dec 3. PMID 21126728